CLINICAL TRIAL: NCT02920242
Title: A Randomized, Double-blind, Parallel Group, Placebo-controlled, Multi-center, Therapeutic Equivalence Study to Compare Rifaximin 200 mg Tablets (Sandoz GmbH) to Xifaxan® 200 mg Tablets (Salix Pharmaceuticals, Inc.) and Placebo in Patients With Travelers' Diarrhea
Brief Title: A Study Comparing Two Rifaximin Tablets in Patients With Travelers' Diarrhea.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated due to low enrollment
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1526 RIF_2
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Results first posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2018-12

CONDITIONS: Travelers' Diarrhea
Keywords: Travelers; diarrhea; rifaximin; equivalence
MeSH Terms: conditions — Diarrhea | interventions — Rifaximin; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rifaximin (Experimental): Patients received Rifaximin 200 mg tablet 3 times per day for 3 days.
  Interventions: Drug: Rifaximin (Sandoz GmbH) tablet
- Xifaxan (Active Comparator): Patients received Xifaxan 200 mg tablet 3 times per day for 3 days.
  Interventions: Drug: Rifaximin (Xifaxan)
- Placebo (Placebo Comparator): Patients received placebo tablet 3 times per day for 3 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin (Sandoz GmbH) tablet — 200 mg tablet administered orally.
  Arms: Rifaximin
Drug: Rifaximin (Xifaxan) — 200 mg tablet administered orally
  Other Names: Xifaxan®
  Arms: Xifaxan
Drug: Placebo — Matching Placebo tablet administered orally
  Arms: Placebo

SUMMARY:
This study compared safety and efficacy of a generic rifaximin tablet to the reference listed drug in the treatment of travelers' diarrhea. Additionally both the generic and reference formulations were tested for superiority against a placebo tablet.

It was planned that 450 patients would be enrolled, but only 28 patients were randomized. Of these, 1 patient discontinued due to failure to meet the inclusion/exclusion criteria. The remaining 27 patients received study drug and 25 patients completed the study.

The study was terminated due to slow enrolment. The final analysis included only safety analysis in the Safety population, due to the low number of randomized patients. No efficacy analysis was performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to read and understood the language of the Informed Consent Form and Patient Information.
* International travelers with a duration of stay in host country long enough to attend schedules visits.
* Affected by naturally acquired acute diarrhea, defined as the passage of at least 3 unformed stools within 24 hours immediately preceding randomization preceding randomization

Exclusion Criteria:

* Hypersensitivity to rifaximin or any of the rifamycin antimicrobial agents or to any of the excipients of the study drug.
* Pregnant, breast feeding or planning pregnancy
* Acute diarrhea for > 72 hours immediately prior to randomization.
* Presence of fever (≥ 100 °F/37.8°C) or hematochezia (blood in stool, noted visually) or clinical findings suggesting moderate or severe dehydration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sandoz Investigative Site, Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rifaximin | Xifaxan | Placebo
Started | 13 | 11 | 4
Safety Set | 12 | 11 | 4
Completed | 11 | 11 | 3
Not Completed | 2 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Did not meet inc./exc. criteria | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics was based on the safety analysis set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rifaximin | Xifaxan | Placebo | Total
Number analyzed (Participants) | 12 | 11 | 4 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.3 (18.27) | 38.2 (18.69) | 35.8 (21.93) | 37.0 (18.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 1 | 13
  Male | 7 | 4 | 3 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 11 | 11 | 4 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure Rate
Description: Clinical cure was defined as either no stools or only formed stools within a 48 hour period and no fever, with or without other enteric symptoms, OR no watery stools or no more than two soft stools passed within a 24 hour period with no fever and no other enteric symptoms except for mild excess gas/flatulence.
Time Frame: study day 5 +/- 1 day
Population: The study was terminated after only 28 patients (6% of planned population) were randomized. In line with the predefined Statistical Analysis Plan (SAP) no efficacy analysis was performed due to low sample size.
Arm/Group | Rifaximin | Xifaxan | Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Time to Last Unformed Stool
Time Frame: within 5 study days
Population: as for outcome 1
Arm/Group | Rifaximin | Xifaxan | Placebo
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Proportion of Patients With Clinical Failure
Time Frame: within 5 study days
Population: as for outcome 1
Arm/Group | Rifaximin | Xifaxan | Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Proportion of Patients With Improvement of Diarrheal Syndrome
Time Frame: within 5 study days
Population: as for outcome 1
Arm/Group | Rifaximin | Xifaxan | Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Number of Unformed Stools
Time Frame: within 5 study days
Population: as for outcome 1
Arm/Group | Rifaximin | Xifaxan | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: The Presence or Absence and Severity of Signs and Symptoms of Enteric Infection
Time Frame: within 5 study days
Population: as for outcome 1
Arm/Group | Rifaximin | Xifaxan | Placebo
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Microbiological Cure Rate
Time Frame: study day 5
Population: as for outcome 1
Arm/Group | Rifaximin | Xifaxan | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to day 5 +/- 1 day
Arm/Group | Rifaximin | Xifaxan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/4
Other Adverse Events (participants affected / at risk) | 2/12 | 5/11 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rifaximin (N=12) | Xifaxan (N=11) | Placebo (N=4)
Lacrimation increased (Eye disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Medication error (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2015-10-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT02920242/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT02920242/SAP_001.pdf